CLINICAL TRIAL: NCT05875129
Title: Intervention for Chronic Insufficient Sleep in Young Adult Cancer Survivors
Brief Title: Device Feasibility and Acceptability to Improve Insomnia in Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: STUDY00006301
Record Dates: First submitted 2023-05-01; First posted 2023-05-25 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Cancer; Insomnia Chronic
MeSH Terms: conditions — Neoplasms; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Through the VAVA (an Amazon Alexa provided as part of the study), participants will verbally provide information about their sleep habits and sleep quality and receive suggestions about how to improve their sleep. Via the VAVA, these interactions will happen through the prototype software More SHEEP (MediaRez LLC). The recommendations provided by the More SHEEP software will be tailored to the individual participant, based on the data provided verbally by each participant. The participant will be asked to engage with the VAVA prototype daily for a 2-week period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental): Participants (N=15) will will be provided with the VAVA prototype along with installation instructions to embed the VAVA within their homes. We provide them with a smart speaker running our intervention, a smart lamp, and a new router. They will be asked to trial the VAVA for a period of 2 weeks, a duration consistent with the primary stage of CBT-I treatment.
  Interventions: Device: VAVA prototype

INTERVENTIONS:
Device: VAVA prototype — Cognitive behavioral therapy for insomnia

SUMMARY:
Sleep disruption is common among young adult cancer survivors for a variety of reasons. Cognitive behavioral therapy for insomnia (CBT-I) has been shown to improve chronic sleep disorders. This project will test the feasibility and acceptability of a new voice-activated virtual assistant (VAVA) device to deliver CBT-I to improve sleep among young adult cancer survivors with chronic sleep disorders.

DETAILED DESCRIPTION:
Sleep is a complex biobehavioral event, impacted by interactions between the individual's physiology as well as their environment. Young adult cancer survivors (YACS; those between 18- 29 years of age) are a growing group of survivors, numbering close to 400,000 in the US. They are among those at highest risk for chronically insufficient sleep due to developmentally normative biological and social factors, compounded by their extensive medical treatment history. Cognitive-behavioral therapy for insomnia (CBT-I) is recommended by the American College of Physicians as gold standard treatment for insomnia disorder and has been successfully adapted for YACS. Fundamental CBT-I strategies can be implemented to change the problematic sleep behaviors that result in insufficient sleep among young adults. However, it is essential that these evidence-based strategies be deployed to be responsive to the specific barriers to sleep for YACS. This feasibility/acceptability study will test the use of an integrated VAVA that offers the opportunity to implement intervention strategies in a way that repeatedly gives YACS the chance to make the right decision with respect to their sleep health in real time.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 29 years old
* history of cancer (any type, any stage)
* chronic sleep loss as evidence by self-report of receiving less sleep than recommended for their age by the National Sleep Foundation for >/= 3 months
* must have an internet router in their primary home that they have access to (can add a second router to for the system to work)

Exclusion Criteria:

* acute medical/psychiatric disorder requiring treatment
* developmental or congenital disorder
* life expectancy <12 months.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2022-07-20 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of device use | 14 days
  Number of days that a participant interacted with the VAVA
Acceptability | 14 days
  Score on satisfaction subscale of Usability, Satisfaction, Ease of use (USE) scale

CONTACTS AND LOCATIONS:
Locations (1):
- MedStar Washington Hospital Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Groninger H, Arem H, Ayangma L, Gong L, Zhou E, Greenberg D. Development of a Voice-Activated Virtual Assistant to Improve Insomnia Among Young Adult Cancer Survivors: Mixed Methods Feasibility and Acceptability Study. JMIR Form Res. 2025 Mar 10;9:e64869. doi: 10.2196/64869. PMID 40063947